CLINICAL TRIAL: NCT02904629
Title: Evaluation of Respecting the Circle of Life on Pregnancy Prevention Outcomes Among American Indian Adolescents
Acronym: TPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6670
Record Dates: First submitted 2016-08-30; First posted 2016-09-19 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Sex; Unprotected Sex; Contraception; Alcohol Use; Drug Use; Pregnancy
MeSH Terms: conditions — Coitus; Unsafe Sex; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RCL Intervention (Experimental): Respecting the Circle of Life (RCL) includes peer-group & youth-parent components. The peer-group component has 8 educational lessons, each lasting 90-120 minutes, delivered to self-selected same-sex peer groups of 8-10 AI teens. RCL lessons are delivered once/day during an 8-day summer basketball camp. The youth-parent component is one educational lesson lasting 90-120 minutes delivered within 3 months after camp to a teen and parent together at home. Total RCL duration is 810-1,080 minutes over 3 months. All 8 days of the camp are "study days," in which RCL youth will receive one lesson each day. The investigators will evaluate RCL's impact on key sexual and reproductive health risk factors at 3-, 9-, 12-, 24-, and 36-month post-intervention follow-up time points.
  Interventions: Behavioral: Respecting the Circle of Life (RCL)
- Control (Other): The control program includes peer-group & youth-parent components. The peer-group component has 8 educational lessons, each lasting 90-120 minutes, delivered to self-selected same-sex peer groups of 8-10 AI teens. Control lessons are delivered once/day during an 8-day summer basketball camp. The youth-parent component is one educational lesson lasting 90-120 minutes delivered within 3 months after camp to a teen and parent together at home. Total control duration is 810-1,080 minutes over 3 months. All 8 days of the camp are "study days," in which control youth will receive one lesson each day. The investigators will evaluate the control program's impact on key sexual and reproductive health risk factors at 3-, 9-, 12-, 24-, and 36-month post-intervention follow-up time points.
  Interventions: Other: Control Program

INTERVENTIONS:
Behavioral: Respecting the Circle of Life (RCL) — Intervention activities will consist of the delivery of RCL: an holistic sexual, reproductive health and teen pregnancy prevention curriculum. RCL was adapted in 2011 from an evidence-based intervention (EBI) for the prevention of HIV/AIDS called "Focus on Youth (FOY) + Informed Parents and Children Together (ImPACT)."
  Arms: RCL Intervention
Other: Control Program — Control activities will consist of the delivery of educational lessons on nutrition, fitness, outdoor recreation, safety, environmental protection and nature.
  Arms: Control

SUMMARY:
The objective of this research study is to evaluate a culturally tailored sexual and reproductive health intervention among American Indian (AI) youth. Specifically, the investigators aim to evaluate the impact of "Respecting the Circle of Life: Mind, Body and Spirit" on knowledge, attitude and behavioral outcomes associated with risk for unprotected sex, sexually transmitted infection (STI) and unintended pregnancy through a randomized controlled trial on the White Mountain Apache (WMA) reservation. The investigators will examine whether the RCL intervention effectively reduces risky sexual behavior among AI adolescents (11-19 years old), with long term goals of reducing teen pregnancy and incidence/prevalence of STIs. The evaluation will focus on well-established intermediate outcomes/risky sexual behaviors that predict long-term impact on teen pregnancy and STI incidence.

DETAILED DESCRIPTION:
The investigators have the following research questions:

Confirmatory Research Question 1: Assess the effectiveness of the RCL intervention, compared to the control condition, on improving knowledge related to reproductive health, pregnancy, contraception and STIs. Outcome Measure 1: Knowledge Score (0-100%): Mean score on a 44-question reproductive and sexual health knowledge survey.

Confirmatory Research Question 2: Assess the effectiveness of the RCL intervention, compared to the control condition, on delaying initiation of sexual activity. Outcome Measure 2: Proportion of participants who report they have ever had sex.

Confirmatory Research Question 3: Assess effectiveness of the RCL intervention, compared to the control condition, on improving condom use self-efficacy. Outcome Measure 3: Condom Use Self-Efficacy Scale (range 1-5): Mean score on a 6-question Likert scale (1-5).

Confirmatory Research Question 4: Assess the effectiveness of the RCL intervention, compared to the control condition, on increasing intention to use a condom at next sex.

Outcome Measure 4: Proportion of participants who report they intend to use a condom at next sex.

Sub-Group Analysis Question 1: Assess the effectiveness of the RCL intervention, compared to the control condition, on increasing reported condom use at last sex among sexually active participants. Sub-Group Analysis Outcome Measure 1: Proportion sexually active participants who report using a condom at last sex.

Sub-Group Analysis Question 2: Assess the effectiveness of the RCL intervention, compared to the control condition, on reducing the number of sexual partners reported by sexually active participants in the past three months. Sub-Group Analysis Outcome Measure 2: Mean number of sexual partners reported in the past three months by sexually active participants.

Sub-Group Analysis Question 3: Assess the effectiveness of the RCL intervention, compared to the control condition, on reducing the number of times sexually active participants reported having sex without a condom in the past three months. Sub-Group Analysis Outcome Measure 3: 1) Proportion of sexually active participants who had sex without a condom in the past three months. 2) Mean number of times reported having sex without a condom in past three months by sexually active participants.

Sub-Group Analysis Question 4: Assess the effectiveness of the RCL intervention, compared to the control condition, on increasing contraceptive use among sexually active participants in the past three months. Sub-Group Analysis Outcome Measure 4: 1) Proportion sexually active participants who had sex without birth control in past three months. 2) Mean number of times reported having sex without birth control in past three months by sexually active participants.

The impact evaluation will also examine two exploratory research questions:

Exploratory Research Question 1: Examine whether the RCL intervention, compared to the control condition, improves parental engagement (communication and monitoring) among teen participants, and whether improved parental engagement is associated with decreased risky sexual behavior among those who are sexually active (as measured by confirmatory research question outcomes).

Exploratory Research Question 2: a) Explore differences in risky sexual behaviors between adolescent participants who do and do not report substance use, and whether the RCL intervention, compared to the control condition, impacts adolescent substance use. b) Examine whether the RCL intervention, compared to the control condition, reduces reported substance use immediately prior to and/or during sex among sexually active participants.

ELIGIBILITY:
Inclusion Criteria:

* American Indian ethnicity
* Membership in the White Mountain Apache community. (Although the investigators anticipate the vast majority of participants will be White Mountain Apache tribal members, study participation is open to all American Indian individuals who live on the Fort Apache Indian Reservation or on/near the border).
* Participants ages 11+ must have parent/legal guardian consent
* Adult participants must sign written informed consent

Exclusion Criteria:

* Inability to participate in full intervention or evaluation (e.g., planned move, residential treatment, etc.)
* Unwilling to be randomized

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1072 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Condom use self efficacy as measured by the Condom Use Self-Efficacy Scale (range 1-5): Mean score on a 6-question Likert scale (1-5) | 3-month, 9-month, 12-month, 24-month, 36-month
  Mean difference in ability to correctly and consistently use condoms, between intervention and control groups at baseline, 3-month, 9-month, 12-month, 24-month, 36-month post-intervention.

SECONDARY OUTCOMES:
Initiation of sexual activity as measured by the proportion of participants who report ever having sex | 3-month, 9-month, 12-month, 24-month, 36-month
  Delayed initiation of sexual activity between intervention and control groups at baseline, 3-month, 9-month, 12-month, 24-month, 36-month post-intervention.
Knowledge of sexual and reproductive health as measured by the mean score on a 44-question reproductive and sexual health knowledge survey | 3-month, 9-month, 12-month, 24-month, 36-month
  Change in knowledge score (range 0-100%) related to sexual and reproductive health, pregnancy and contraception between intervention and control groups at between baseline, 3-month, 9-month, 12-month, 24-month, 36-month post-intervention.
Condom use intention as measured by the proportion of participants who report they intend to use a condom at next sex | 3-month, 9-month, 12-month, 24-month, 36-month
  Change in intention to use a condom at next sex, between intervention and control groups at baseline, 3-month, 9-month, 12-month, 24-month, 36-month post-intervention

OTHER OUTCOMES:
Condom use at last sex as measured by the proportion of sexually active participants who report using a condom at last sex | 3-month, 9-month, 12-month, 24-month, 36-month
  Condom use at last sex among sexually active participants between intervention and controls groups at baseline, 3-month, 9-month, 12-month, 24-month, 36-month post-intervention
Number of sexual partners as measured by the mean number of sexual partners reported in the past 3 months | 3-month, 9-month, 12-month, 24-month, 36-month
  Number of sexual partners among sexually active participants, between intervention and control groups at baseline, 3-month, 9-month, 12-month, 24-month, 36-month post-intervention
Sexual activity without using a condom as measured by the proportion of participants who had sex without a condom in the past 3 months and the mean number of times reported having sex without a condom in the past 3 months | 3-month, 9-month, 12-month, 24-month, 36-month
  Sexual activity without using a condom among sexually active participants between intervention and control groups at baseline, 3-month, 9-month, 12-month, 24-month, 36-month post-intervention.
Contraceptive use as measured by the proportion of sexually active participants who had sex without birth control in the past 3 months and the mean number of times reported having sex without birth control in past 3 months | 3-month
  Contraceptive use among sexually active participants in past three months, by sexually active participants, between intervention and control groups at 3-month post-intervention.
Parental engagement as measured by the Parent-Adolescent Communication Scale: (Mean Score on 39-item Likert Scale) and the Parental Monitoring Scale: (Mean Score on a 6-item Likert Scale) | 3-month, 9-month, 12-month, 24-month, 36-month
  Parental engagement with youth participants (communication and monitoring) between intervention and control groups at baseline, 3-month, 9-month, 12-month, 24-month, 36-month post-intervention.
Risky sexual behaviors as measured by the proportion who report having unprotected sex in the past 3 months among participants who use alcohol and drugs | 3-month
  Risky sexual behavior in last 3 months among participants who use alcohol and drugs, between intervention and control groups.
Substance use during sex as measured by the proportion who use alcohol or drugs immediately prior to and/or during sex | 3-month, 9-month, 12-month, 24-month, 36-month
  Substance use immediately prior and/or during sex, among sexually active participants between intervention and control groups at baseline, 3-month, 9-month, 12-month, 24-month and 36-month post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barlow, PhD, Study Director — Center for American Indian Health; Lauren Tingey, PhD, Principal Investigator — Center for American Indian Health
Locations (1):
- Johns Hopkins Center for American Indian Health, Whiteriver, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The funding body (Office of Adolescent Health) requires sharing of de-identified data.

REFERENCES:
- [Derived] Tingey L, Chambers R, Patel H, Littlepage S, Lee S, Lee A, Susan D, Melgar L, Slimp A, Rosenstock S. Prevention of Sexually Transmitted Diseases and Pregnancy Prevention Among Native American Youths: A Randomized Controlled Trial, 2016-2018. Am J Public Health. 2021 Oct;111(10):1874-1884. doi: 10.2105/AJPH.2021.306447. Epub 2021 Sep 16. PMID 34529503
- [Derived] Tingey L, Chambers R, Goklish N, Larzelere F, Lee A, Suttle R, Rosenstock S, Lake K, Barlow A. Rigorous evaluation of a pregnancy prevention program for American Indian youth and adolescents: study protocol for a randomized controlled trial. Trials. 2017 Feb 27;18(1):89. doi: 10.1186/s13063-017-1842-6. PMID 28241775